CLINICAL TRIAL: NCT00167375
Title: Testing the Nocturnal Sleep Latency Profile in Primary Insomnia
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: American Academy of Sleep Medicine (Other); Sumitomo Pharma America, Inc. (Industry)
Other Study IDs: NSLP1; 27-CA-04
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Primary Insomnia; Sleep Initiation and Maintenance Disorders
Keywords: Insomnia; polysomnography; sleep onset; time series analysis
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone; Behavior Therapy

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: eszopiclone 3 mg qHS
Behavioral: General cognitive/behavioral interventions for insomnia

SUMMARY:
This study tests a new kind of sleep study in which subjects are awakened 2 times after initially going to sleep. The study focuses on the EEG signal process as a person goes to sleep. The general hypothesis is that the signal properties are stable from night to night during baseline studies, and are different between controls and patients with primary insomnia. The primary insomnia patients then go on to have about 2 weeks of an insomnia intervention. Then the new kind of study is repeated in the patients. The controls only are examined in baseline studies.

DETAILED DESCRIPTION:
Patients are carefully screened to have DSM primary insomnia, and do not have another disorder than may cause a sleep disturbance. After a 2-week baseline period, the subjects undergo a screening sleep study to rule out sleep apnea and periodic limb movement disorder. Then they undergo the NSLP procedure. In that procedure, there pre-bedtime EEG recordings and questionnaire responses taken. Then at a planned time, the subjects go to bed and try to sleep while there EEG signals are recorded. After the first and second sleep cycles, they are awakened for one minute, then asked to return to sleep. In the morning additional recordings and questionnaire responses are obtained. Two nights later they repeat a baseline NSLP procedure. The controls then end their participation. The Patients then receive an open treatment with eszopiclone and behavioral treatments so that their insomnia may improve. After 2 weeks intervention, the patients complete one NLSP night. The goal of the study is to see if there can be data to support the idea that the sleep onset process might harbor a sign of primary insomnia that could be used for the development of a better medical model of primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Primary Insomnia (N = 12) Age & Gender matched Healthy controls (N = 12)

Exclusion Criteria:

* Unstable Medical illness No other Sleep disorder BMI > 35, AHI > 10, PLM Index > 10, Ferritin < 50. Unable to communicate in English

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2005-01; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas E Moul, M.D., M.P.H, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States